CLINICAL TRIAL: NCT01686997
Title: 'Effect of Long biLiopancrEatic Limb lenGth in lAparoscopic Roux-eN-Y Gastric Bypass on Weight Loss and Comorbidities in Patients With Morbid obEsity: a Prospective Randomized Control Trial'
Brief Title: Effect of Long Biliopancreatic Limb RYGB on Weight Loss and Comorbidities
Acronym: Elegance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Elegance01
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Morbid Obesity
Keywords: Bariatric surgery; Roux-en-Y Gastric Bypass
MeSH Terms: conditions — Obesity, Morbid | interventions — Gastric Bypass

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Primairy long biliopancreatic limb RYGB (Active Comparator): Roux limb 75 cm and Biliopancreatic Limb 150 cm
  Interventions: Procedure: Roux-en-Y Gastric Bypass
- Redo Long biliopancreatic limb RYGB (Active Comparator): Roux limb 75 cm and Biliopancreatic limb 150 cm
  Interventions: Procedure: Roux-en-Y Gastric Bypass
- Primairy standard RYGB (Active Comparator): Roux limb 150 cm and Biliopancreatic limb 75 cm
  Interventions: Procedure: Roux-en-Y Gastric Bypass
- Redo standard RYGB (Active Comparator): Roux limb 150 cm and Biliopancreatic limb 75 cm
  Interventions: Procedure: Roux-en-Y Gastric Bypass

INTERVENTIONS:
Procedure: Roux-en-Y Gastric Bypass

SUMMARY:
Morbid obesity is an increasing medical problem in the western countries. It's related to comorbidities as diabetes mellitus, hypertension, OSAS, arthrosis and hypercholesterolemia. The Roux-en-Y Gastric Bypass (RYGB) is an effective surgical therapy for morbidly obese patients. A part of these patients will have disappointing results, and have weight regain on the long term. Some studies show more weight reduction by increasing the biliopancreatic limb in patients with morbid obesity.

The objective of this study is to investigate the effect of variations in the length of biliopancreatic limb on weight reduction in morbidly obese patients undergoing RYGB-surgery. We hypothesize that longer biliopancreatic limb results in more weight reduction.

The study design is a prospective, randomized control trial. The patients will be randomized in 2 groups: a standard RYGB (short biliopancreatic limb) and long biliopancreatic limb RYGB.

ELIGIBILITY:
Inclusion Criteria:

Patient eligible for bariatric surgery according Fried guidelines

Primary Gastric bypass

* BMI 35 - 40 with a comorbidity
* or BMI > 40

Redo- operation

* medical history: gastric sleeve/ mason / gastric band
* all BMI levels

Exclusion Criteria:

* Exclusion criteria for bariatric surgery (Fried Guidelines)
* Patients with language problems that interveins to follow medical advises
* Genetic diseases that intervens to follow medical advises
* Chronic bowel diseases
* Nephrologic (MDRD <30) of liver diseases (AST/ALT more than twice the norm)
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2012-07; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Weight reduction | 2 years
  excess weight loss (%EWL)

SECONDARY OUTCOMES:
Decrease in comorbidities | 2 years
  diabetes mellitus, hypertension, hypercholesterolemia, arthrosis
Quality of life | 2 years
  SF-36 and BAROS
Complications and re-operations | 2 years
  bleeding, wound infections, intra-abdominal abcess, anastomosis leakage, vitamine deficiencies

CONTACTS AND LOCATIONS:
Overall Officials: F.J. Berends, MD, PhD, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate Hospital, Arnhem, Netherlands

REFERENCES:
- [Derived] Homan J, Boerboom A, Aarts E, Dogan K, van Laarhoven C, Janssen I, Berends F. A Longer Biliopancreatic Limb in Roux-en-Y Gastric Bypass Improves Weight Loss in the First Years After Surgery: Results of a Randomized Controlled Trial. Obes Surg. 2018 Dec;28(12):3744-3755. doi: 10.1007/s11695-018-3421-7. PMID 30073496